CLINICAL TRIAL: NCT05240677
Title: Value of Esophageogastroduodenscopy in Assessment of Chronic Kidney Disease Patients With Iron Deficiency Anemia Without Gastrointestinal Symptoms
Brief Title: Endoscopy in CKD With Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walid Ahmed Ragab Abdelhamid (Other Government)
Responsible Party: Sponsor-Investigator, Walid Ahmed Ragab Abdelhamid, Lecturer internal medicine, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9145/2-2-2022
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases; Iron-Deficiency Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): Chronic kidney diseases patients with iron deficiency anemia and eGFR ≥ 60 ml/min/1.73 m2
  Interventions: Procedure: Upper GIT endoscopy
- Group 2 (Experimental): Chronic kidney diseases patients with iron deficiency anemia and eGFR < 60 ml/min/1.73 m2.
  Interventions: Procedure: Upper GIT endoscopy

INTERVENTIONS:
Procedure: Upper GIT endoscopy — Upper gastrointestinal endoscpy for all participants and gastric biopsy for histopathological examination for suspicious lesions

SUMMARY:
Iron deficiency anemia is very common in CKD patients. Data about gastrointestinal lesions in Arab patients are insufficient.

DETAILED DESCRIPTION:
Iron deficiency anemia without gastrointestinal symptoms needs to be assessed in patients with chronic kidney disease.

ELIGIBILITY:
* Patients with eGFR is less than 60 ml/m/1.73 m2.
* Patients with iron deficiency anemia.
* Absence of gastrointestinal symptoms.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of upper gastrointestinal endoscopic findings In chronic kidney disease patients with iron deficiency anemia | 6 months
  Detect rate of upper GIT lesions in asymptomatic CKD patients with iron deficiency anemia using endoscopy followed by biopsy and histopathological examination

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No